CLINICAL TRIAL: NCT07380373
Title: Comparative Analysis of Salivary and Bronchoalveolar Lavage IL-6 and TNF-α as Biomazrkers in Pediatric Acute Respiratory Distress Syndrome
Brief Title: Comparative Analysis of Salivary and Bronchoalveolar Lavage IL-6 and TNF-α as Biomarkers in Pediatric Acute Respiratory Distress Syndrome
Status: Enrolling by invitation | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MD88/2025
Record Dates: First submitted 2025-12-20; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-04

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
Keywords: ARDS; Salivary biomarkers; IL-6; TNF alfa; BAL biomarkers
MeSH Terms: conditions — Acute Lung Injury | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bronchoscopy — Comparison between levels of inflammatory markers in both BAL &salivary secretions

SUMMARY:
The aim of this study is to determine the degree of agreement in cytokines level measured through BAL and those measured through salivary glands excretion.

and to compare the validity of cytokines in BAL versus salivary secretion in predicting the stage of ARDS and disease outcome in term of mortality, disease progression and length of stay.

DETAILED DESCRIPTION:
• BAL will be performed by the attending pediatric intensivist in pediatric intensive care unit as part of standard care for ARDS management and Saliva samples will be collected non-invasively using sterile collection devices IL6 and TNF alfa will measured in both samples and compared to each other

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Pediatric Acute Respiratory Distress Syndrome (ARDS)
* Age range: 1 month to 18 years
* Requirement for invasive mechanical ventilation
* Availability of salivary and bronchoalveolar lavage (BAL) samples within 24 hours of ARDS diagnosis
* Informed consent obtained from parent or legal guardian

Exclusion Criteria:

* Pre-existing chronic lung disease (e.g., cystic fibrosis, bronchopulmonary dysplasia)
* Known immunodeficiency or current immunosuppressive therapy
* Active malignancy or receipt of chemotherapy within the past 6 months
* Severe congenital anomalies incompatible with survival
* Refusal or inability to obtain informed consent

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of pediatric patients diagnosed with mild to moderate acute respiratory distress syndrome (ARDS) who are admitted to the pediatric intensive care unit (PICU) and on mechanical ventilation to decrease the hazards of bronchoscopy on sever patients with ARDS
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Agreement between BAL and salivary cytokine levels | Within 24 hours of ARDS diagnosis
  Degree of agreement between cytokine concentrations measured in bronchoalveolar lavage (BAL) fluid and salivary gland secretions collected simultaneously, assessed using intraclass correlation coefficients and Bland-Altman analysis.

SECONDARY OUTCOMES:
Prediction of ARDS severity by cytokine levels | First 48-72 hours
  Ability of BAL and salivary cytokine levels to predict ARDS severity according to established criteria.
Association of cytokine levels with in-hospital mortality | Through the study completion ( anaverage one year)
  Relationship between cytokine concentrations and all-cause in-hospital mortality.
Association of cytokine levels with disease progression | Through the study completion of average one year
  Relationship between cytokine levels and worsening ARDS severity or escalation of respiratory support.
Association of cytokine levels with length of hospital stay | Through the study completion ( an average one year)
  Relationship between cytokine concentrations and length of hospital stay.
Comparative predictive performance of BAL versus salivary cytokines | Through a study completion of average one year
  Comparison of BAL and salivary cytokines in predicting ARDS severity, mortality, disease progression, and length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tarekahmed Abdelgawad, Study Director — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the primary research team